CLINICAL TRIAL: NCT04020809
Title: Neoadjuvant Atezolizumab in Patients With Non-Metastatic Resectable High-Risk Cutaneous Melanoma
Brief Title: Neoadjuvant Atezolizumab in Cutaneous Melanoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Nestor Esnaola, Professor of Surgery, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML41440
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cutaneous Melanoma
Keywords: atezolizumab; neoadjuvant; cutaneous melanoma
MeSH Terms: conditions — Melanoma | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atezolizumab (Experimental): Atezolizumab will be administered as 1200 mg intravenously on Day 1 every 3 weeks for 2 cycles.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Anti-PD-L1 monoclonal antibody
  Other Names: Tecentriq

SUMMARY:
The purpose of this research study is to see whether using atezolizumab before surgery is safe and does not cause side effects that delay surgery in participants with cutaneous melanoma that has not spread to other areas of the body (non-metastatic) and can be removed by surgery (resectable) but has a higher risk of coming back after surgery (high-risk).

DETAILED DESCRIPTION:
The purpose of this study is to test the safety of using atezolizumab before surgery in participants with cutaneous melanoma that has not spread to other areas of the body (non-metastatic) and can be removed by surgery (resectable) but has a higher risk of coming back after surgery (high-risk). Cutaneous melanoma in its earliest stages before it has spread to other areas of the body can usually be cured with surgery alone. Unfortunately, some cutaneous melanomas have a greater likelihood of coming back after surgery. Your immune system is normally your body's first defense against threats like cancer. But sometimes cancer cells produce signals that allow them to hide from attack by the immune system. One such signal is called programmed cell death-ligand 1 (PD-L1). Atezolizumab is a drug that blocks PD-L1. By blocking PD-L1, atezolizumab may boost your immune system to keep your cutaneous melanoma from coming back after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Female or male.
* Age ≥18 years at time of signing informed consent form.
* Ability to comply with the trial protocol, in the investigator's judgment.
* Histologically confirmed cutaneous melanoma with pathological evidence of residual disease in place.
* Clinically non-metastatic (stage I-II) disease.
* Technically resectable disease (no significant vascular, neural, or bony involvement and potential to safely achieve R0 resection) per the treating surgical oncologist.
* High-risk disease (clinical stage IA-IIC disease meeting criteria for sentinel lymph node biopsy as per the National Comprehensive Cancer Network guidelines [clinical stage IB-IIC (i.e., T1b-T4bN0M0) OR clinical stage IA (T1aN0M0) with high risk denoted by T1a with greater than or equal to 2 mitoses per mm2 OR lymphovascular invasion OR their combination]).
* Treatment-naïve.
* Eastern Cooperative Oncology Group performance status of 0-2.
* Adequate hematologic and end-organ function.
* Negative human immunodeficiency virus (HIV) test at screening, with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥200/µL, and have an undetectable viral load.
* Negative hepatitis B surface antigen test at screening.
* Willing to provide biopsy and blood specimens as required by the trial.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of <1% per year during the treatment period and for 5 months after the final dose of trial treatment. Women must also refrain from donating eggs during this same period.

Exclusion Criteria:

* Anal melanoma, vaginal melanoma, mucosal melanoma, or melanoma of soft parts.
* History of leptomeningeal disease.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).
* Uncontrolled or symptomatic hypercalcemia.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis scan.
* Active tuberculosis.
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of trial treatment, unstable arrhythmia, or unstable angina.
* Major surgical procedure within 4 weeks prior to initiation of trial treatment.
* Severe infection within 4 weeks prior to initiation of trial treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Treatment with therapeutic oral or intravenous antibiotics within 2 weeks prior to initiation of trial treatment.
* Prior allogeneic stem cell or solid organ transplantation.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of trial treatment, or anticipation of need for such a vaccine during trial treatment or within 5 months after the final dose of trial treatment.
* Current treatment with anti-viral therapy for hepatitis B virus.
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-cytotoxic T lymphocyte-associated antigen-4, anti-programmed cell death-1, and anti-PD-L1 therapeutic antibodies.
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin-2 within 4 weeks or 5 half-lives of the drug [whichever is longer]) prior to initiation of trial treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-alpha agents) within 2 weeks prior to initiation of trial treatment, or anticipation of need for systemic immunosuppressive medication during trial treatment.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* Current use of anticoagulants at therapeutic levels.
* Prior active malignancy within the previous 2 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or cervical cancer in place that have undergone potentially curative therapy.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation.
* Pregnancy or breastfeeding, or intention of becoming pregnant during trial treatment or within 5 months after the final dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants completing neoadjuvant atezolizumab | 63 months
  Determine the number of participants who complete the 2 neoadjuvant doses of atezolizumab without any extended treatment-related delay (defined as >80 days from Cycle 1 to date of surgical resection)
Number of participants with treatment-related adverse events | 63 months
  Determine the number of participants with treatment-related adverse events, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events v5.0

SECONDARY OUTCOMES:
Pathological response rate in primary tumor and sentinel lymph node(s) | 63 months
  Determine the pathological response rate in primary tumor and sentinel lymph node(s) of neoadjuvant atezolizumab
Two-year recurrence-free survival (RFS) rate | 63 months
  Determine the 2-year RFS rate of neoadjuvant atezolizumab
Two-year overall survival (OS) rate | 63 months
  Determine the 2-year OS rate of neoadjuvant atezolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Esnaola, M.D., Principal Investigator — Houston Methodist Cancer Center
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No